CLINICAL TRIAL: NCT01825499
Title: Vermont Oxford Network Very Low Birth Weight Database of Infants <=1500 Grams or <=29 Weeks Gestational Age At Birth
Brief Title: Vermont Oxford Network Very Low Birth Weight Database
Acronym: VON VLBW
Status: Recruiting | Type: Observational
Sponsor: Vermont Oxford Network (Network)
Responsible Party: Sponsor
Other Study IDs: VON001
Record Dates: First submitted 2013-03-27; First posted 2013-04-05 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Neonatology
Keywords: Birth weight; Gestational age; Very low birth weight; Infant; Neonatal
MeSH Terms: conditions — Birth Weight | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Very low birth weight infants: Infants <=1500 g or <=29 weeks gestational age admitted to Vermont Oxford Network member centers within 28 days of birth
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry

SUMMARY:
Vermont Oxford Network maintains a database for live born infants <=1500 grams or <=29 weeks gestational age who are born at participating hospitals or admitted to them within 28 days of birth, regardless of where in the hospital the infant receives care.

DETAILED DESCRIPTION:
The Database collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The information collected is not specific to a disease or treatment. The data collected includes information on:

* Demographics of mother and infant
* Mother's health, labor and delivery
* Infant's health upon admission, procedures and interventions, and medical outcomes

These data are used to: provide member centers with reporting for use in quality improvement; examine associations between baseline characteristics, treatments, and outcomes; and track trends in incidences of disease and effectiveness of therapies.

ELIGIBILITY:
Inclusion Criteria:

* Any infant who is born alive and whose birth weight is <=1500 grams or <=29 weeks 6 days gestational age (inclusive) who is born at or admitted to a Vermont Oxford Network member center within 28 days of life without having first gone home, regardless of the where the infant receives care

Exclusion Criteria:

* Stillborn infants
* Infants discharged home prior to admission to a member center
* Infants admitted after 28 days

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who are <=1500 grams birth weight or <=29 weeks gestational age and who are admitted to Vermont Oxford Network member centers within 28 days of birth without first going home
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 1990-01; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Registry of baseline and outcome data for VLBW infants with data collected in a uniform manner | up to 1 year
  Data items include infant and maternal characteristics, delivery room interventions, respiratory care and outcomes, surgeries, infections, other serious complications, and length of stay. Time frames for data collection include: characteristics of birth; at day 28; and at discharge. Tracking ends at discharge home (including for infants transferred out) or at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Horbar, MD, Study Chair — Vermont Oxford Network
Locations (1):
- Vermont Oxford Network, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prakalapakorn SG, Greenberg L, Edwards EM, Ehret DEY. Trends in Retinopathy of Prematurity Screening and Treatment: 2008-2018. Pediatrics. 2021 Jun;147(6):e2020039966. doi: 10.1542/peds.2020-039966. Epub 2021 May 11. PMID 33975923
- [Background] Jensen EA, Edwards EM, Greenberg LT, Soll RF, Ehret DEY, Horbar JD. Severity of Bronchopulmonary Dysplasia Among Very Preterm Infants in the United States. Pediatrics. 2021 Jul;148(1):e2020030007. doi: 10.1542/peds.2020-030007. Epub 2021 Jun 2. PMID 34078747
- [Background] Edwards EM, Greenberg LT, Profit J, Draper D, Helkey D, Horbar JD. Quality of Care in US NICUs by Race and Ethnicity. Pediatrics. 2021 Aug;148(2):e2020037622. doi: 10.1542/peds.2020-037622. Epub 2021 Jul 22. PMID 34301773
- [Background] Flannery DD, Edwards EM, Puopolo KM, Horbar JD. Early-Onset Sepsis Among Very Preterm Infants. Pediatrics. 2021 Oct;148(4):e2021052456. doi: 10.1542/peds.2021-052456. Epub 2021 Sep 7. PMID 34493539
- [Background] Boghossian NS, Geraci M, Edwards EM, Horbar JD. Changes in hospital quality at hospitals serving black and hispanic newborns below 30 weeks' gestation. J Perinatol. 2022 Feb;42(2):187-194. doi: 10.1038/s41372-021-01222-3. Epub 2021 Oct 2. PMID 34601491
- [Background] Runte KE, Flyer JN, Edwards EM, Soll RF, Horbar JD, Yeager SB. Variation of Patent Ductus Arteriosus Treatment in Very Low Birth Weight Infants. Pediatrics. 2021 Nov;148(5):e2021052874. doi: 10.1542/peds.2021-052874. Epub 2021 Oct 21. PMID 34675131
- [Background] Edwards EM, Greenberg LT, Ehret DEY, Soll RF, Lanzieri TM, Horbar JD. STORCH Infections Among Very Low Birth Weight and Preterm Infants: 2018-2020. Pediatrics. 2022 Jan 1;149(1):e2021053655. doi: 10.1542/peds.2021-053655. No abstract available. PMID 35104887
- [Background] Keefe G, Culbreath K, Edwards EM, Morrow KA, Soll RF, Modi BP, Horbar JD, Jaksic T. Current outcomes of infants with esophageal atresia and tracheoesophageal fistula: A multicenter analysis. J Pediatr Surg. 2022 Jun;57(6):970-974. doi: 10.1016/j.jpedsurg.2022.01.060. Epub 2022 Feb 14. PMID 35300859
- [Background] Culbreath K, Keefe G, Edwards EM, Morrow KA, Soll RF, Jaksic T, Horbar JD, Modi BP. Morbidity associated with laparotomy-confirmed spontaneous intestinal perforation: A prospective multicenter analysis. J Pediatr Surg. 2022 Jun;57(6):981-985. doi: 10.1016/j.jpedsurg.2022.01.058. Epub 2022 Feb 14. PMID 35287964
- [Background] Salazar EG, Handley SC, Greenberg LT, Edwards EM, Lorch SA. Measuring quality of care in moderate and late preterm infants. J Perinatol. 2022 Oct;42(10):1294-1300. doi: 10.1038/s41372-022-01377-7. Epub 2022 Mar 30. PMID 35354940
- [Background] Boghossian NS, Greenberg LT, Edwards EM, Horbar JD. Transfer Patterns of Very Low Birth Weight Infants for Convalescent Care. Pediatrics. 2022 Jun 1;149(6):e2021054866. doi: 10.1542/peds.2021-054866. PMID 35588188
- [Background] Culbreath K, Knell J, Keefe G, Nes E, Han SM, Edwards EM, Morrow KA, Soll RF, Jaksic T, Horbar JD, Modi BP. Impact of concomitant necrotizing enterocolitis on mortality in very low birth weight infants with intraventricular hemorrhage. J Perinatol. 2023 Jan;43(1):91-96. doi: 10.1038/s41372-022-01434-1. Epub 2022 Jun 17. PMID 35715599
- [Background] Handley SC, Salazar EG, Greenberg LT, Foglia EE, Lorch SA, Edwards EM. Variation and Temporal Trends in Delivery Room Management of Moderate and Late Preterm Infants. Pediatrics. 2022 Aug 1;150(2):e2021055994. doi: 10.1542/peds.2021-055994. PMID 35851607
- [Background] Mangiza M, Ehret DEY, Edwards EM, Rhoda N, Tooke L. Morbidity and mortality in small for gestational age very preterm infants in a middle-income country. Front Pediatr. 2022 Aug 9;10:915796. doi: 10.3389/fped.2022.915796. eCollection 2022. PMID 36016879
- [Background] Flannery DD, Edwards EM, Coggins SA, Horbar JD, Puopolo KM. Late-Onset Sepsis Among Very Preterm Infants. Pediatrics. 2022 Dec 1;150(6):e2022058813. doi: 10.1542/peds.2022-058813. PMID 36366916
- [Background] Fraiman YS, Edwards EM, Horbar JD, Mercier CE, Soll RF, Litt JS. Racial Inequity in High-Risk Infant Follow-Up Among Extremely Low Birth Weight Infants. Pediatrics. 2023 Feb 1;151(2):e2022057865. doi: 10.1542/peds.2022-057865. PMID 36594226
- [Background] Salazar EG, Handley SC, Greenberg LT, Edwards EM, Lorch SA. Association Between Neonatal Intensive Care Unit Type and Quality of Care in Moderate and Late Preterm Infants. JAMA Pediatr. 2023 Mar 1;177(3):278-285. doi: 10.1001/jamapediatrics.2022.5213. PMID 36648939
- [Background] Edwards EM, Greenberg LT, Horbar JD, Gagliardi L, Adams M, Berger A, Leitao S, Luyt K, Ehret DEY, Rogowski JA. Discharge Age and Weight for Very Preterm Infants in Six Countries: 2012-2020. Neonatology. 2023;120(2):208-216. doi: 10.1159/000528013. Epub 2023 Jan 17. PMID 36649689
- [Background] Coggins SA, Edwards EM, Flannery DD, Gerber JS, Horbar JD, Puopolo KM. Serratia Infection Epidemiology Among Very Preterm Infants in the Neonatal Intensive Care Unit. Pediatr Infect Dis J. 2023 Feb 1;42(2):152-158. doi: 10.1097/INF.0000000000003736. Epub 2022 Nov 2. PMID 36638403
- [Background] Boghossian NS, Geraci M, Phibbs CS, Lorch SA, Edwards EM, Horbar JD. Trends in Resources for Neonatal Intensive Care at Delivery Hospitals for Infants Born Younger Than 30 Weeks' Gestation, 2009-2020. JAMA Netw Open. 2023 May 1;6(5):e2312107. doi: 10.1001/jamanetworkopen.2023.12107. PMID 37145593
- [Background] Agha L, Staiger D, Brown C, Soll RF, Horbar JD, Edwards EM. Association of Hospital Adoption of Probiotics With Outcomes Among Neonates With Very Low Birth Weight. JAMA Health Forum. 2023 May 5;4(5):e230960. doi: 10.1001/jamahealthforum.2023.0960. PMID 37171798
- [Background] Frade Garcia A, Edwards EM, de Andrade Lopes JM, Tooke L, Assenga E, Ehret DEY, Hansen A. Neonatal Admission Temperature in Middle- and High-Income Countries. Pediatrics. 2023 Sep 1;152(3):e2023061607. doi: 10.1542/peds.2023-061607. PMID 37589082
- [Background] Rogowski J, Greenberg L, Edwards E, Ehret D, Horbar J. Horizontally integrated health systems and neonatal intensive care unit (NICU) care for very preterm infants. Health Aff Sch. 2023 Sep 11;1(3):qxad042. doi: 10.1093/haschl/qxad042. eCollection 2023 Sep. PMID 38756675
- [Background] Culbreath K, Keefe G, Nes E, Edwards EM, Knell J, Morrow KA, Soll RF, Jaksic T, Horbar JD, Modi BP. Association between neurodevelopmental outcomes and concomitant presence of NEC and IVH in extremely low birth weight infants. J Perinatol. 2024 Jan;44(1):108-115. doi: 10.1038/s41372-023-01780-8. Epub 2023 Sep 21. PMID 37735208
- [Background] Munoz FA, Carter EH, Edwards EM, Jerome M, Litt JS. Does faster weight trajectory lead to improved neurodevelopmental outcomes in ELBW infants with bronchopulmonary dysplasia? J Perinatol. 2024 Feb;44(2):301-306. doi: 10.1038/s41372-023-01808-z. Epub 2023 Oct 28. PMID 37898685
- [Background] Horbar JD, Greenberg LT, Buzas JS, Ehret DEY, Soll RF, Edwards EM. Trends in Mortality and Morbidities for Infants Born 24 to 28 Weeks in the US: 1997-2021. Pediatrics. 2024 Jan 1;153(1):e2023064153. doi: 10.1542/peds.2023-064153. PMID 38053449
- [Background] Handley SC, Salazar EG, Kunz SN, Lorch SA, Edwards EM. Transfer Patterns Among Infants Born at 28 to 34 Weeks' Gestation. Pediatrics. 2024 Jan 1;153(2):e2023063118. doi: 10.1542/peds.2023-063118. PMID 38268423
- [Background] Nes E, Chugh PV, Keefe G, Culbreath K, Morrow KA, Ehret DEY, Soll RF, Horbar JD, Harting MT, Lally KP, Modi BP, Jaksic T, Edwards EM. Predictors of Mortality in Very Low Birth Weight Neonates With Congenital Diaphragmatic Hernia. J Pediatr Surg. 2024 May;59(5):818-824. doi: 10.1016/j.jpedsurg.2024.01.032. Epub 2024 Feb 1. PMID 38368194
- [Background] Chugh PV, Nes E, Culbreath K, Keefe G, Edwards EM, Morrow KA, Ehret D, Soll RF, Modi BP, Horbar JD, Jaksic T. Comparing Healthcare Needs in Extremely Low Birth Weight Infants With NEC and Spontaneous Intestinal Perforation. J Pediatr Surg. 2024 Sep;59(9):1759-1764. doi: 10.1016/j.jpedsurg.2024.03.006. Epub 2024 Mar 16. PMID 38561308
- [Background] Edwards EM, Ehret DEY, Horbar JD. Potentially Better Practices for Follow Through in Neonatal Intensive Care Units. Pediatrics. 2024 Jul 1;154(1):e2023065530. doi: 10.1542/peds.2023-065530. PMID 38872618
- [Background] Leahy BF, Edwards EM, Ehret DEY, Soll RF, Yeager SB, Flyer JN. Transcatheter and Surgical Ductus Arteriosus Closure in Very Low Birth Weight Infants: 2018-2022. Pediatrics. 2024 Aug 1;154(2):e2024065905. doi: 10.1542/peds.2024-065905. PMID 39005106
- [Background] Edwards EM, Ehret DEY, Soll RF, Horbar JD. Survival of Infants Born at 22 to 25 Weeks' Gestation Receiving Care in the NICU: 2020-2022. Pediatrics. 2024 Oct 1;154(4):e2024065963. doi: 10.1542/peds.2024-065963. PMID 39323403
- [Background] Lake ET, Staiger D, Horbar J, Cheung R, Kenny MJ, Patrick T, Rogowski JA. Association between hospital recognition for nursing excellence and outcomes of very low-birth-weight infants. JAMA. 2012 Apr 25;307(16):1709-16. doi: 10.1001/jama.2012.504. PMID 22535856
- [Background] Fitzgibbons SC, Ching Y, Yu D, Carpenter J, Kenny M, Weldon C, Lillehei C, Valim C, Horbar JD, Jaksic T. Mortality of necrotizing enterocolitis expressed by birth weight categories. J Pediatr Surg. 2009 Jun;44(6):1072-5; discussion 1075-6. doi: 10.1016/j.jpedsurg.2009.02.013. PMID 19524719
- [Background] Zupancic JA, Richardson DK, Horbar JD, Carpenter JH, Lee SK, Escobar GJ; Vermont Oxford Network SNAP Pilot Project Participants. Revalidation of the Score for Neonatal Acute Physiology in the Vermont Oxford Network. Pediatrics. 2007 Jan;119(1):e156-63. doi: 10.1542/peds.2005-2957. Epub 2006 Dec 11. PMID 17158947
- [Background] Walsh MC, Yao Q, Horbar JD, Carpenter JH, Lee SK, Ohlsson A. Changes in the use of postnatal steroids for bronchopulmonary dysplasia in 3 large neonatal networks. Pediatrics. 2006 Nov;118(5):e1328-35. doi: 10.1542/peds.2006-0359. PMID 17079534
- [Background] Morales LS, Staiger D, Horbar JD, Carpenter J, Kenny M, Geppert J, Rogowski J. Mortality among very low-birthweight infants in hospitals serving minority populations. Am J Public Health. 2005 Dec;95(12):2206-12. doi: 10.2105/AJPH.2004.046730. PMID 16304133
- [Background] Rogowski JA, Staiger DO, Horbar JD. Variations in the quality of care for very-low-birthweight infants: implications for policy. Health Aff (Millwood). 2004 Sep-Oct;23(5):88-97. doi: 10.1377/hlthaff.23.5.88. PMID 15371373
- [Background] Lucey JF, Rowan CA, Shiono P, Wilkinson AR, Kilpatrick S, Payne NR, Horbar J, Carpenter J, Rogowski J, Soll RF. Fetal infants: the fate of 4172 infants with birth weights of 401 to 500 grams--the Vermont Oxford Network experience (1996-2000). Pediatrics. 2004 Jun;113(6):1559-66. doi: 10.1542/peds.113.6.1559. PMID 15173474
- [Background] Rogowski JA, Horbar JD, Staiger DO, Kenny M, Carpenter J, Geppert J. Indirect vs direct hospital quality indicators for very low-birth-weight infants. JAMA. 2004 Jan 14;291(2):202-9. doi: 10.1001/jama.291.2.202. PMID 14722146
- [Background] Suresh GK, Horbar JD, Kenny M, Carpenter JH; Vermont Oxford Network. Major birth defects in very low birth weight infants in the Vermont Oxford Network. J Pediatr. 2001 Sep;139(3):366-73. doi: 10.1067/mpd.2001.117072. PMID 11562615
- [Background] Horbar JD, Badger GJ, Lewit EM, Rogowski J, Shiono PH. Hospital and patient characteristics associated with variation in 28-day mortality rates for very low birth weight infants. Vermont Oxford Network. Pediatrics. 1997 Feb;99(2):149-56. doi: 10.1542/peds.99.2.149. PMID 9024438
- [Background] Horbar JD. Increasing use of antenatal corticosteroid therapy between 1990 and 1993 in Vermont Oxford Network. J Perinatol. 1997 Jul-Aug;17(4):309-13. PMID 9280098
- [Background] De Nisi G, Berti M, Malossi R, Pederzini F, Pedrotti A, Valente A. Comparison of neonatal intensive care: Trento area versus Vermont Oxford Network. Ital J Pediatr. 2009 Mar 14;35(1):5. doi: 10.1186/1824-7288-35-5. PMID 19490662
- [Background] Hull MA, Fisher JG, Gutierrez IM, Jones BA, Kang KH, Kenny M, Zurakowski D, Modi BP, Horbar JD, Jaksic T. Mortality and management of surgical necrotizing enterocolitis in very low birth weight neonates: a prospective cohort study. J Am Coll Surg. 2014 Jun;218(6):1148-55. doi: 10.1016/j.jamcollsurg.2013.11.015. Epub 2013 Nov 27. PMID 24468227
- [Background] Fisher JG, Jones BA, Gutierrez IM, Hull MA, Kang KH, Kenny M, Zurakowski D, Modi BP, Horbar JD, Jaksic T. Mortality associated with laparotomy-confirmed neonatal spontaneous intestinal perforation: a prospective 5-year multicenter analysis. J Pediatr Surg. 2014 Aug;49(8):1215-9. doi: 10.1016/j.jpedsurg.2013.11.051. Epub 2013 Nov 15. PMID 25092079
- [Background] Lake ET, Staiger D, Horbar J, Kenny MJ, Patrick T, Rogowski JA. Disparities in perinatal quality outcomes for very low birth weight infants in neonatal intensive care. Health Serv Res. 2015 Apr;50(2):374-97. doi: 10.1111/1475-6773.12225. Epub 2014 Sep 22. PMID 25250882
- [Background] Fisher JG, Bairdain S, Sparks EA, Khan FA, Archer JM, Kenny M, Edwards EM, Soll RF, Modi BP, Yeager S, Horbar JD, Jaksic T. Serious congenital heart disease and necrotizing enterocolitis in very low birth weight neonates. J Am Coll Surg. 2015 Jun;220(6):1018-1026.e14. doi: 10.1016/j.jamcollsurg.2014.11.026. Epub 2014 Dec 9. PMID 25868405
- [Background] Fullerton BS, Sparks EA, Morrow KA, Edwards EM, Soll RF, Jaksic T, Horbar JD, Modi BP. Hospital transfers and patterns of mortality in very low birth weight neonates with surgical necrotizing enterocolitis. J Pediatr Surg. 2016 Jun;51(6):932-5. doi: 10.1016/j.jpedsurg.2016.02.051. Epub 2016 Mar 3. PMID 27230800
- [Background] McBride CA, Bernstein IM, Badger GJ, Horbar JD, Soll RF. The effect of maternal hypertension on mortality in infants 22, 29weeks gestation. Pregnancy Hypertens. 2015 Oct;5(4):362-6. doi: 10.1016/j.preghy.2015.10.002. Epub 2015 Oct 27. PMID 26597755
- [Background] Hallowell SG, Rogowski JA, Spatz DL, Hanlon AL, Kenny M, Lake ET. Factors associated with infant feeding of human milk at discharge from neonatal intensive care: Cross-sectional analysis of nurse survey and infant outcomes data. Int J Nurs Stud. 2016 Jan;53:190-203. doi: 10.1016/j.ijnurstu.2015.09.016. Epub 2015 Oct 9. PMID 26518107
- [Background] Horbar JD, Ehrenkranz RA, Badger GJ, Edwards EM, Morrow KA, Soll RF, Buzas JS, Bertino E, Gagliardi L, Bellu R. Weight Growth Velocity and Postnatal Growth Failure in Infants 501 to 1500 Grams: 2000-2013. Pediatrics. 2015 Jul;136(1):e84-92. doi: 10.1542/peds.2015-0129. PMID 26101360
- [Background] Horbar JD, Edwards EM, Greenberg LT, Morrow KA, Soll RF, Buus-Frank ME, Buzas JS. Variation in Performance of Neonatal Intensive Care Units in the United States. JAMA Pediatr. 2017 Mar 6;171(3):e164396. doi: 10.1001/jamapediatrics.2016.4396. Epub 2017 Mar 6. PMID 28068438
- [Background] Fullerton BS, Hong CR, Velazco CS, Mercier CE, Morrow KA, Edwards EM, Ferrelli KR, Soll RF, Modi BP, Horbar JD, Jaksic T. Severe neurodevelopmental disability and healthcare needs among survivors of medical and surgical necrotizing enterocolitis: A prospective cohort study. J Pediatr Surg. 2017 Oct 12:S0022-3468(17)30651-6. doi: 10.1016/j.jpedsurg.2017.10.029. Online ahead of print. PMID 29079317
- [Background] Boghossian NS, Geraci M, Edwards EM, Morrow KA, Horbar JD. Anthropometric Charts for Infants Born Between 22 and 29 Weeks' Gestation. Pediatrics. 2016 Dec;138(6):e20161641. doi: 10.1542/peds.2016-1641. Epub 2016 Nov 18. PMID 27940694
- [Background] Horbar JD, Edwards EM, Greenberg LT, Profit J, Draper D, Helkey D, Lorch SA, Lee HC, Phibbs CS, Rogowski J, Gould JB, Firebaugh G. Racial Segregation and Inequality in the Neonatal Intensive Care Unit for Very Low-Birth-Weight and Very Preterm Infants. JAMA Pediatr. 2019 May 1;173(5):455-461. doi: 10.1001/jamapediatrics.2019.0241. PMID 30907924
- [Background] Belfort MB, Edwards EM, Greenberg LT, Parker MG, Ehret DY, Horbar JD. Diet, weight gain, and head growth in hospitalized US very preterm infants: a 10-year observational study. Am J Clin Nutr. 2019 May 1;109(5):1373-1379. doi: 10.1093/ajcn/nqz008. PMID 30997514
- [Background] Smith BJ, Flyer JN, Edwards EM, Soll RF, Horbar JD, Yeager SB. Outcomes for Ectopia Cordis. J Pediatr. 2020 Jan;216:67-72. doi: 10.1016/j.jpeds.2019.09.014. Epub 2019 Oct 24. PMID 31668886
- [Background] Han SM, Watters KF, Hong CR, Edwards EM, Knell J, Morrow KA, Soll RF, Jaksic T, Horbar JD, Modi BP. Tracheostomy in Very Low Birth Weight Infants: A Prospective Multicenter Study. Pediatrics. 2020 Mar;145(3):e20192371. doi: 10.1542/peds.2019-2371. Epub 2020 Feb 25. PMID 32098788
- [Background] Gray MM, Edwards EM, Ehret DEY, Brei BK, Greenberg LT, Umoren RA, Ringer S, Horbar J. Resuscitation Opportunities for Fellows of Very Low Birth Weight Infants in the Vermont Oxford Network. Pediatrics. 2020 Jul;146(1):e20193641. doi: 10.1542/peds.2019-3641. Epub 2020 Jun 12. PMID 32532791
- See also: Public website with links to manuals and forms, additional articles, research guidelines — http://public.vtoxford.org